CLINICAL TRIAL: NCT03880903
Title: A Prospective Study on the Use of Hypertonic Saline Inhalation in Acute Bronchiolitis in Children
Brief Title: Hypertonic Saline Inhalation in Acute Bronchiolitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MASamoael, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-03

CONDITIONS: Acute Bronchiolitis
MeSH Terms: interventions — Saline Solution; Albuterol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline with bronchdilator (Experimental): will recieve treatment with nebulized brochodilator(salbutamol) and normal saline every 4 to 6 hours
  Interventions: Drug: normal saline and salbutamol
- hypertonic saline with bronchodilator (Experimental): will recieve treatment with nebulized bronchodilator(salbutamol) and hypertonic saline every 4 to 6 hours
  Interventions: Drug: hypertonic saline and salbutamol
- hypertonic saline only (Experimental): will recieve treatment with nebulized hypertonic saline 3% in adose of 4 ml every 4 to 6 hours
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: normal saline and salbutamol — patients will recieve treatment with nebulized salbutamol and normal saline every 4 to 6 in hours
  Arms: normal saline with bronchdilator
Drug: hypertonic saline and salbutamol — patients will recieve treatment with nebulized salbutamol and hypertonic saline 3% in adose of 4ml every 4 to 6 hours
  Arms: hypertonic saline with bronchodilator
Drug: Hypertonic saline — patients will recieve treatment with nebulized hypertonic saline 3% in adose of 4ml every 4 to 6 hours
  Arms: hypertonic saline only

SUMMARY:
Acute bronchiolitis is a viral infection that occurs in children most commonly in the first 2 years of life and is characterized by respiratory symptoms, resulting in wheezing and/or crackles upon auscultation. It is usually a self limiting illness. However, this condition may be associated with several severe complications, such as apnea,respiratory failure, or secondary bacterial infection

DETAILED DESCRIPTION:
Acute bronchiolitis is a viral infection that occurs in children most commonly in the first 2 years of life and is characterized by respiratory symptoms, resulting in wheezing and/or crackles upon auscultation. It is usually a self limiting illness. However, this condition may be associated with several severe complications, such as apnea,respiratory failure, or secondary bacterial infection. Bronchiolitis is a significant cause of respiratory disease worldwide. according to the World Health Organization bullet in, an estimated 150 million new cases occur annually; 11-20 million (7-13%) of these cases are severe enough to require hospital admission. Worldwide, 95% of all cases occur in developing countries. Typically, initial clinical manifestations include upper respiratory tract symptoms such as cough, nasal congestion, and low-grade fever lasting 1 to 3 days, followed by expiratory wheezing, nasal flaring, fine crackles, oxygen saturation on presentation<94%, tachypnea, increased work of breathing, use of accessory muscles, and retractions in some patients. The need for hospitalization depends on the presence of respiratory symptoms (degree of retractions, increased respiratory effort, decreased oxygen saturation), cyanosis, restlessness or lethargy, and underlying disease states, including apnea. Since no definitive antiviral therapy exists for most causes of bronchiolitis, management of these infants should be directed toward symptomatic relief and maintenance of hydration and oxygenation. One medication that has demonstrated promising results in the management of acute bronchiolitis is nebulized hypertonic saline , Its hyperosmolarity helps to absorb water from the mucosal and submucosal space, thereby increasing mucociliary function by clearing fluids accumulated in the airway and mucus plugs in the lungs. Hypertonic saline can also induce cough to help enhance mucus clearance. The American Academy Of Pediatrics guidelines recommend administration of hypertonic saline in hospitalized bronchiolitis patients. The most common dosage studied is hypertonic saline 3% 4 mL per dose inhaled by nebulizer every 4 to 6 hours, which may take ≥24 hours to work and is typically continued while the child is hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* infants less than 24 months of age with adiagnosis of acute bronchiolitis

Exclusion Criteria:

* other infants and children above 24 months of age
* patients with other diseases than acute bronchiolitis

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | 24 hours
  time taken to discharge or ready to be discharged

REFERENCES:
- [Result] Teshome G, Gattu R, Brown R. Acute bronchiolitis. Pediatr Clin North Am. 2013 Oct;60(5):1019-34. doi: 10.1016/j.pcl.2013.06.005. Epub 2013 Jul 24. PMID 24093893
- [Result] Smyth RL, Openshaw PJ. Bronchiolitis. Lancet. 2006 Jul 22;368(9532):312-22. doi: 10.1016/S0140-6736(06)69077-6. PMID 16860701
- [Result] Rudan I, Tomaskovic L, Boschi-Pinto C, Campbell H; WHO Child Health Epidemiology Reference Group. Global estimate of the incidence of clinical pneumonia among children under five years of age. Bull World Health Organ. 2004 Dec;82(12):895-903. Epub 2005 Jan 5. PMID 15654403
- [Result] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768